CLINICAL TRIAL: NCT05982847
Title: National Blood Pressure Screening in Children to Optimise Clinical Management of Paediatric Hypertension in South Africa
Brief Title: National Blood Pressure Screening in Children to Improve Paediatric Healthcare in South Africa
Status: Recruiting | Type: Observational
Sponsor: North-West University, South Africa (Other)
Collaborators: Medical Research Council, South Africa (Other); University of Cape Town (Other); University of Limpopo (Other); Walter Sisulu University (Other); University of KwaZulu (Other); Red Cross War Memorial Childrens Hospital (Other); University of Witwatersrand, South Africa (Other); University of Zurich (Other); Groote Schuur Hospital (Unknown); Nelson Mandela Metropolitan University (Other); Chris Hani Baragwanath Academic Hospital (Other); University of the Free State (Unknown)
Responsible Party: Principal Investigator, Ruan Kruger, Professor, North-West University, South Africa
Other Study IDs: REC 4/23/03/22
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Obesity, Adolescent; Obesity, Childhood
Keywords: Adiposity; Blood Pressure; Cardiovascular Diseases; Health Knowledge, Attitudes, Practice; Lifestyle Factors
MeSH Terms: conditions — Hypertension; Pediatric Obesity; Obesity; Cardiovascular Diseases; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boys
  Interventions: Diagnostic Test: Blood pressure screening
- Girls
  Interventions: Diagnostic Test: Blood pressure screening

INTERVENTIONS:
Diagnostic Test: Blood pressure screening — Blood pressure and anthropometric measurements will be performed in children and adolescents between ages 5-18 years to develop South African nomograms that will aid in the development of clinical practice guidelines to optimise hypertension care in South Africa youth.
  Other Names: Anthropometric measurements

SUMMARY:
The Childhood Hypertension Consortium of South Africa (CHCSA) was established to foster relationships between the healthcare sector and schools through community engagement and outreach as well as contributing to the decolonization of normative paediatric blood pressure reference values. To date, there has been no nation-wide project in South Africa to determine nationally representative normal blood pressure reference values, nor to estimate the true prevalence of hypertension in the paediatric population of the country. This study will provide critical information on the understanding of blood pressure and hypertension in children, especially of African ancestry. Not only will this effort contribute to the development of the first nationally representative normal reference values of blood pressure but will also benefit healthcare providers in the sector with a clear guideline on the management of high blood pressure in children as developed by experts working with these challenges daily.

DETAILED DESCRIPTION:
Rationale: Currently there exist no nationally representative set of normative reference values for blood pressure and anthropometry in South African children, while clinicians rely on European and US reference values. The latter seems inappropriate in the South African setting, especially considering the lack of data available in African ancestry normative data.

Objectives: The investigators aim to development the first nationally representative normal reference values of blood pressure and anthropometry in children, to develop scientific evidence-based hypertension guidelines in the paediatric population of South Africa.

Methods: The target population for this study includes 5 to under 18 years school-aged (all school quintiles) children in South Africa from all provinces in the country selected in a randomized manner and to ensure generalizability.

Population: A sample of 22 464 (81% Black African; 9% Coloured; 8% White and 2% Indian/Asian) will be required to enable computation of reference values for each age and sex across urban, peri-urban and rural settings in all provinces.

Time frame: The study will recruit and collect data over a period of five years.

Expected outcomes: The investigators expect that normative blood pressure in children (ages above 5 and under 18 years) will differ from currently accepted international thresholds. The investigators will engage in the communities to optimise awareness and care of high blood pressure and its comorbidities. Recommendations will be made to the National Department of Health regarding blood pressure measurement/screening for hypertension in children at the local clinic in the Road to Health booklet. The investigators will also develop the first clinical practice guidelines for the management of hypertension in children in South Africa in collaboration with hypertension societies.

ELIGIBILITY:
Inclusion Criteria:

* All children between ages 5-<18 years
* All children with voluntary assent/consent and parent's permission

Exclusion Criteria:

* circumstances interfere with the participant's ability to give informed consent (diminished understanding or comprehension, or any language barriers that may pose potential risk in participation under false expectations)
* randomly selected children who choose not to participate (lack of assent/consent), even if parent's permission was received,
* conditions that interfere with a patient's ability to follow study guidelines, e.g., the use of drugs, alcohol or tobacco products
* ages >18 years or under 5 years
* Children will be excluded from the analysis for the determination of normative reference values for blood pressure and anthropometry if taking certain concomitant medication(s) that may affect their blood pressure, or any underlying disease e.g., chronic kidney disease, chronic heart disease etc. that may raise blood pressure.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The target population for this study includes 5 to under 18 years school-aged children in South Africa from all provinces in the country selected in a randomized manner and to ensure generalizability. All South African public ordinary schools are categorised into five groups, called quintiles, largely for purposes of the allocation of financial resources from government. Quintile one is the lowest socioeconomic quintile, while quintile five is the highest. In addition, lower quintile schools are mostly rural and/or peri-urban. Participants will be drawn from quintile 1-5 schools and those in more remote areas will be reached via mobile fieldwork teams. A sample of 22 464 (81% Black African; 9% Coloured; 8% White and 2% Indian/Asian) will be required to enable computation of reference values for each age and sex across urban and rural settings in all provinces.
Sampling Method: Probability Sample
Enrollment: 22464 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
To determine and compute nationally representative normative reference values for blood pressure in children | Through study completion, an average of 1 year
  To date there are no national normative blood pressure reference values for children in South Africa. Normative values used by clinicians are those extrapolated from studies on blood pressure done in the USA and Europe and these may not be truly representative of normative values of blood pressure in South Africa. This study aims to address this issue, because children can be misdiagnosed for high blood pressure based on the wrong normative values.
To determine and compute nationally representative normative reference values for blood pressure in children | Through study completion, an average of 1 year
  Overweight and obesity classification according to the World Health Organisation percentiles for childhood obesity only include a small sample size from less than five African countries, therefore the underrepresentation of children of African ancestry will be addressed by this study.
To develop clinical practice guidelines for the management of childhood hypertension in South Africa | Through study completion, an average of 1 year
  The findings of this study will help develop clinically relevant guidelines for the management of hypertension in children between 5 and 18 years of age based on local normative values, as well as to improve cost and availability of anti-hypertensive agents for children and adolescents.

CONTACTS AND LOCATIONS:
Locations (11):
- South Africa (10):
  - Walter Sisulu University, Mthatha, Eastern Cape
  - Nelson Mandela Metropolitan University, Port Elizabeth, Eastern Cape
  - University of the Free State, Bloemfontein, Free State
  - University of the Witwatersrand, Johannesburg, Gauteng
  - University of KwaZulu-Natal, Durban, KwaZulu-Natal
  - University of Limpopo, Polokwane, Limpopo
  - Hypertension in Africa Research Team (HART), North-West University, Potchefstroom, North West
  - Red Cross War Memorial Children Hospital, Cape Town, Western Cape
  - South African Medical Research Council, Cape Town, Western Cape
  - University of Cape Town, Cape Town, Western Cape
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The national data will be first collated to develop the nomograms for blood pressure and anthropometric measurements. The data will be made available upon reasonable request from the principal investigator(s) after publication of the nomograms findings.